CLINICAL TRIAL: NCT04195295
Title: Regeneration of Intrabony Defects With Nano Hydroxyapatite Graft, Derived From Egg Shell Along With Periosteum as Barrier Membrane Under Magnification - An Interventional Study
Brief Title: Regeneration of Intrabony Defects With Nano Hydroxyapatite Graft, and Periosteum as Barrier Membrane Under Magnification
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Principal Investigator, Dr Prabhuji MLV, Professor and HOD, Krishnadevaraya College of Dental Sciences & Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02_D012_102133
Record Dates: First submitted 2019-12-06; First posted 2019-12-11 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Intrabony Periodontal Defect

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- periosteal membrane and egg shell graft (Experimental): Egg shell derived nano hydroxyapatite (EnHA) as regenerative graft material and periosteal pedicle as barrier membrane.
  Interventions: Procedure: Regeneration of Intrabony Defects with Nano Hydroxyapatite Graft, Derived from Egg Shell along with Periosteum as Barrier Membrane
- only egg shell graft (Experimental): Only Egg shell derived nano hydroxyapatite (EnHA) as graft material.
  Interventions: Procedure: Regeneration of intrabony defects using Egg shell derived nano hydroxyapatite (EnHA) as regenerative graft material
- open flap debridement (Active Comparator): open flap debridement procedure only.
  Interventions: Procedure: Open flap debridement procedure in intrabony defects.

INTERVENTIONS:
Procedure: Regeneration of Intrabony Defects with Nano Hydroxyapatite Graft, Derived from Egg Shell along with Periosteum as Barrier Membrane — * In group A, the full thickness mucoperiosteal flap will be elevated, which will be extended apically to expose sufficient amount of periosteum.
  * Periosteal membrane will be separated from the full thickness mucoperiosteal flap and released by one vertical incision mesially and one horizontal incision apically.
  * Posteriorly, the periosteum remained attached with the mucoperiosteal flap, so that blood supply could be maintained in the reflected periosteum.
  * Then the graft material will be packed into the defect.
  * Then periosteal membrane will be turned over the intrabony defect in such a way that the defect was completely covered by the periosteal membrane
  Arms: periosteal membrane and egg shell graft
Procedure: Regeneration of intrabony defects using Egg shell derived nano hydroxyapatite (EnHA) as regenerative graft material — Full thickness mucoperiosteal flap will be raised and Vertical releasing incisions are used if necessary for better access to the surgical site. Then EnHA graft material will be placed into the defect before suturing the mucoperiosteal flap.
  Arms: only egg shell graft
Procedure: Open flap debridement procedure in intrabony defects. — full thickness mucoperiosteal flap will be raised, entire granulation tissue will be removed from the defects, the pocket epithelium was curetted from the inner surface of the flap, and the roots were thoroughly scaled and planed by means of manual and ultrasonic instruments. Then the operative area will be irrigated with sterile saline. After that, the mucoperiosteal flaps will be sutured.
  Arms: open flap debridement

SUMMARY:
The prospective study is a interventional study to evaluate and compare the effectiveness of periosteal pedicle as grafting technique and egg shell derived nano hydroxyapatite as regenerative graft material for regeneration of intrabony defects.

DETAILED DESCRIPTION:
30 Patients visiting the outpatient Department of Periodontology Krishnadevaraya College of Dental Sciences and Hospital, Bangalore will be enrolled for 6 month folllow up study based on the inclusion and exclusion criteria. Patients age ranged from 25 to 55 years. Patients with chronic periodontitis, with presence of intrabony defects with ≥6mm probing depth (PD), 2 or 3 wall defects are included in the study.

The patients are allocated to three goups through computer generated randomisation as:

Group A (n=10) - Egg shell derived nano hydroxyapatite (EnHA) graft and periosteal pedicle as barrier membrane.

Group B (n=10) - Only EnHA as graft. Group C (n=10) - An open flap debridement procedure only.

ELIGIBILITY:
Inclusion Criteria:

1. Patients within the age group of 25 to 55 years.
2. Patients with chronic periodontitis, with presence of intrabony defects with ≥6mm probing depth (PD), 2 or 3 wall defects as detected on CBCT.
3. Gingival biotype >1.5mm
4. Systemically healthy subjects.
5. Patients who are compliant.
6. Patients who had not received any periodontal treatment in the last six months.

Exclusion Criteria:

1. Pregnant and Lactating females.
2. Aggressive periodontitis.
3. Presence of pulpal or periapical involvement.
4. Patients with known systemic diseases and conditions precluding any elective surgery.
5. Patients who were smokers.
6. Teeth with poor prognosis.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Bone defect fill and density | 6 months
  bone defect fill and bone density will be measured pre operatively and post operatively using CBCT

SECONDARY OUTCOMES:
Probing pocket depth | 6 months
  probing pocket depth is measured using UNC 15 probe pre operatively and post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rashmi P, MDS, Principal Investigator — Krishnadevaraya College of Dental Sciences
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No